CLINICAL TRIAL: NCT00711386
Title: A Double-Blind, Randomized, Placebo-Controlled, Repeat Dose Escalation Study to Investigate the Safety, Tolerability and Pharmacokinetics of GSK706769 in Healthy Male and Female Subjects
Brief Title: GSK706769 Repeat Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CRR111382
Record Dates: First submitted 2008-07-03; First posted 2008-07-08 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: pharmacokinetics; CCR5; Healthy volunteers; GSK706769
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort A (Experimental): 50mg dose once daily for 7 days.
  Interventions: Drug: GSK706769; Other: Placebo
- Cohort B (Experimental): 100mg dose once daily for 8 days.
  Interventions: Drug: GSK706769; Other: Placebo
- Cohort C (Experimental): 200mg dose once daily for 8 days.
  Interventions: Drug: GSK706769; Other: Placebo
- Cohort D (Experimental): 400mg dose once daily for 7 days.
  Interventions: Drug: GSK706769; Other: Placebo

INTERVENTIONS:
Drug: GSK706769 — 50mg, 100mg, 200mg, or 400mg
Other: Placebo — Placebo

SUMMARY:
To determine safety, tolerability and Pharmacokinetics of GSK706769

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 50 years of age.
* A female subject is eligible to participate if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who:
* Is pre-menopausal with a documented bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries) or hysterectomy, or
* Is post-menopausal defined as 12 months of spontaneous amenorrhea. A follicle stimulating hormone (FSH) level will be performed to confirm a post-menopausal status. For this study, FSH levels > 40 mlU/ml is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt, HRT should be discontinued for 2 weeks and then the subject rescreened, as HRT can suppress FSH.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 14 days after the last dose of study medication.
* Body weight ³ 50 kg for men and ³ 45 kg for women and BMI within the range 18.5-31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as:
* An average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.

History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation. This includes subjects with a history of known or suspected sulfa related hypersensitivity.

* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol. If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* Has a history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* Consumption of grapefruit or grapefruit juice from 7 days prior to the first dose of study medication until the last pharmacokinetic sample.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy should be excluded.
* Exclusion criteria for screening as per protocol.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting surgery or percutaneous transluminal coronary angioplasty or any clinically significant cardiac disease.
* History/evidence of clinically significant pulmonary disease. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), direct bilirubin or creatinine values greater than the upper limit of normal. A single repeat is allowed for eligibility determination.
* History of significant renal or hepatic diseases.
* Exclusion Criteria for 24-Hour Screening Holter as per protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-05-16 (Actual); Primary Completion 2008-09-12 (Actual); Study Completion 2008-09-12 (Actual)

PRIMARY OUTCOMES:
GSK706769 safety parameters: the number of adverse events | From Day 1 to the follow up visit. Approximately 19 Days.
GSK706769 safety parameters: clinical safety labs from predose values. | From Day 1 to the follow up visit. Approximately 19 Days.
  Change from baseline values in clinical chemistry, hematology and urinalysis.
GSK706769 safety parameters: vital signs (blood pressure and heart rate) from predose values | From Day 1 to the follow up visit. Approximately 19 days.
  Change from baseline values
GSK706769 safety parameters: electrocardiogram (ECG) intervals, ECG rhythm, and ECG axis from predose values. | From Day 1 to the follow up visit. Approximately 19 days.
  Change from baseline values
GSK706769 and GSK1996847 (metabolite) pharmacokinetic parameters following single dose administration on Day 1, when possible | Day 7 or 8
  Area under the plasma concentration time curve (AUC(0-infinity), AUC(0-24)), maximum observed concentration (Cmax), time to maximum observed concentration (tmax), concentration at 24 hours post dose (C24), terminal half-life (t1/2), absorption lag time (tlag), apparent clearance (CL/F), metabolite-to-parent molar ratios for AUC(0-t) and Cmax; and following last repeat administration on Day 7 or 8: AUC(0-infinity), concentration at end of dosing interval (Ctau), Cmax, tlag, tmax, t1/2, and CL/F, metabolite-to-parent molar ratios for AUC(0-tau) and Cmax on Day 7 or 8.

SECONDARY OUTCOMES:
Plasma AUC(0-t), AUC(0-infinity), and CL/F of midazolam, with and without GSK706769 co-administration | Day -1 and Day 8
Plasma AUC(0-t) and Cmax of GSK706769 and GSK1996847 | on Day 7 (fasted) and Day 8 (fed).
GSK706769 and GSK1996847 Day 7 AUC(0-t), Cmax, and Ct compared to Day 1 AUC(0-24), Cmax, and C24, respectively, to estimate accumulation ratios (R) for AUC, Cmax, and Ct. | Day 1 and Day 7
Pre-morning dose concentrations (Ct) on Day 3 through 7 to assess the achievement of steady state of GSK706769 and GSK1996847 following repeat administration. | Day 3 through 7
Day 7 AUC(0-t), Cmax and Ct of GSK706769 and GSK1996847 at different doses for the assessment of dose proportionality. | Day -1 and Day 7

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Madison, Wisconsin, United States

REFERENCES:
- See also: Results for study CRR111382 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/CRR111382?search=study&search_terms=CRR111382#rs